CLINICAL TRIAL: NCT03647605
Title: Pilot Study: Feasibility, Usability and Safety Assessment of VR Mind and VR Mind+ Intervention
Brief Title: Pilot Study: VR Mind and VR Mind+ Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tomorrow Sp. z o.o. (Industry)
Collaborators: National Center for Research and Development, Poland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: POIR.01.01.01-00-0636/16-00
Record Dates: First submitted 2018-06-18; First posted 2018-08-27 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Social Phobia
Keywords: vr; virtual reality; social phobia; vret; virtual reality exposure therapy
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR Mind (Experimental): Two VR Mind sessions using experimental virtual reality scenarios. During these two sessions, participants will be exposed to virtual reality environment, for 2 x 10 min each session.
  Interventions: Behavioral: VR Mind

INTERVENTIONS:
Behavioral: VR Mind — Two VR Mind sessions using virtual reality scenarios concerning social situations in which social phobics are prone to experience anxiety. The pilot study will consist of two scenarios: "Public Speaking in Lecture Hall" and "Telephoning in Public". Two sessions are planned, each containing two expositions to virtual reality environment, each lasting 10 minutes.

SUMMARY:
The aim of the pilot study is feasibility, usability and safety assessment of VR Mind intervention. In particular the subject of assessment will be:

* the length of the laboratory session utilizing virtual reality exposure (feasibility),
* the ergonomics and ease of use for both patients and system operators (usability),
* the frequency of side effect occurrence as a result of virtual reality exposure (ie. Vertigo) (safety).

The results pilot study will be used in the designing a clinical trial aimed for testing efficacy and safety of VR Mind intervention.

DETAILED DESCRIPTION:
In this study, investigators will test the software developed by Tomorrow Sp. z o. o., named VR Mind. The software utilizes the concept of virtual reality exposure therapy to treat social anxiety disorder. The pilot investigators will be tested for the feasibility, usability and safety of the system in order to obtain information useful in further designs for the clinical trial. The research consists of four laboratory sessions. The first and the last session will be dedicated to participant assessment. During the second and third session the virtual reality scenarios (2 x 10 minutes for each session) will be presented to participants. The participants will be playing a role of someone who is giving a speech (Public speaking scenario) and someone who is speaking on a phone in public (Telephoning in public scenario).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-50 y.o.
2. Confirmed DSM-IV-TR criteria for Social Anxiety Disorder (SAD).
3. Signing informed consent

Exclusion Criteria:

1. Occurrence of SAD symptoms inconsistent with DSM-IV-TR criteria and with psychiatric interview (SCID-I; Structured Clinical Interview)
2. Occurrence and/or recognition:

   1. psychosis,
   2. bipolar disorder,
   3. mental retardation
3. Exclusion based on interview:

   1. pregnancy,
   2. drug addiction,
   3. alcohol addiction,
   4. participating in the experimental session while intoxicated
   5. (current) neurological treatment of chronic disease of central nervous system,
   6. epilepsy,
   7. paroxysmal vertigo,
   8. presence of suicidal thoughts , tendencies or attempts,
   9. participant is taking drugs from benzodiazepine group, other sedatives, narcotic drugs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Feasibility_1: Number of participants, who have completed 4 laboratory sessions within 2 weeks. | At the end of 4th laboratory session within 2 weeks
  Number of participants, who have completed 4 laboratory sessions within 2 weeks.
Feasibility_2: Number of virtual reality exposure sessions completed in predefined time. | At the end of 2nd and 3th laboratory session within 2 weeks
  Number of virtual reality exposure sessions completed in predefined time.
Usability_ 3: immersion, perceived reality and engagement | At the end of 2 and 3 laboratory session within 2 weeks
  3 items with 7-point scale, where 1 is "Totally agree" and 7 "Totally disagree":
  1. The virtual reality immersed me in all aspects (Immersion),
  2. The virtual reality resembled true experiences (Reality),
  3. The virtual reality was engaging (Engagement).
Safety_1: occurrence and severity of simulator sickness | During 2nd and 3th laboratory session within 2 weeks
  Simulator sickness is expected adverse effect of the VR. Hence, the Simulator Sickness Questionnaire (SSQ; Kennedy, Lane, Berbaum, Lilienthal, 1993) will be administered as a primary outcome measure to evaluate safety of the VR intervention.
  Total SSQ score equal to or higher than 10 will be used as a preliminary cut-off for simulator sickness (Balk et al., 2013). Individual scores will be corrected for baseline (pre-VR) symptom severity. Only items with a pre-VR - post-VR increase will contribute to a final SSQ score. All post-intervention SSQ scores >10 will be analyzed further for its association with study drop-outs and other intervention required. The adverse effect will be classified as:
  * mild (no intervention required, all VR sessions completed),
  * moderate (any intervention needed, e.g. session termination),
  * severe (hospitalization required),
  * life-threatening / death. Any unexpected adverse effects will be recorded by a physician and classified as described above.

OTHER OUTCOMES:
Clinical Global Impression | During 1st and 4th session within 2 weeks
  Clinical Global Impression (Guy, 1976) - is a single item, 7 point scale used by clinicians to asses the severity of illness, where 1 is labeled as "Normal, not at all ill" and 7 is labeled as "Among the most extremely ill patients".
Patient Global Impression | During 1st and 4th session within 2 weeks
  Patient Global Impression - is a single item, 4 point scale used by patients to asses their impression of severity of their illness and quality of their functioning in everyday life, where 1 is labeled as "Normal" and 4 is labeled as "Severe".
Liebowitz Social Anxiety Scale | During 1st and 4th session within 2 weeks
  Liebowitz Social Anxiety Scale (LSAS; Leibowitz, 1987)
  The scale is composed of 24 items, depicting various social situations. For each item, participants assess their fear (from 1 - "No fear" to 4 - "Severe") and avoidance (from 1 - "Never" to 4 - "Usually").
  LSAS has 3 scores, summing the results for particular items - fear (0-72), avoidance (0-72) and total score (0-144).
Beck Depression Inventory | During 1st and 4th session within 2 weeks
Subjective Units of Distress | During 2nd and 3th session within 2 weeks
  Subjective Units of Distress (SUD)
  SUD is a subjective measure of perceived fear in certain situation. The scale range is from 0 ("Totally relaxed) to 100 ("Highest distress/fear/anxiety/discomfort that you have ever felt").

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Mierzejewski, prof, Principal Investigator — Tomorrow Sp. z o.o.
Locations (1):
- Instytut Psychiatrii i Neurologii, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided